CLINICAL TRIAL: NCT02150109
Title: User Performance of the Karajishi Contour Blood Glucose Monitoring System (ISO/FDA Study)
Brief Title: Evaluation of an Karajishi Contour Investigational Blood Glucose Monitoring System (ISO/FDA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-2014-002-01
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Persons With Diabetes (Experimental): Untrained subjects WITH Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Interventions: Device: Subjects WITH Diabetes Use Karajishi Contour BGMS
- Persons With and Without Diabetes (Experimental): Untrained subjects WITH/WITHOUT Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Interventions: Device: Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS

INTERVENTIONS:
Device: Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS — Untrained subjects WITH and WITHOUT diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood (and study staff tested subject fingerstick blood) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
  Arms: Persons With and Without Diabetes
Device: Subjects WITH Diabetes Use Karajishi Contour BGMS — Untrained subjects WITH diabetes use the Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood (and study staff tested subject fingerstick blood) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
  Arms: Persons With Diabetes

SUMMARY:
The purpose of this study was to determine if untrained persons with diabetes and without diabetes could operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid blood glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual, or neurological impairments that would make the person unable to perform testing with the BGM
* Previously participated in a BG monitor study using the Karajishi Contour BGMS (or used a Bayer Contour meter)
* Work for a medical laboratory, hospital, or other clinical setting that involves training on and clinical use of blood glucose monitors
* Work for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

General enrollment guidelines:

* Most subjects will be persons with type 1 or type 2 diabetes
* At least 10% of subjects with diabetes will have type 1 diabetes
* Approximately 10% of subjects will be persons without diabetes
* At least 60% of subjects will be younger than age 65

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Klaff, MD, Principal Investigator — Rainier Clinical Research Center; Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Rainier Clinical Research Center, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Persons With and Without Diabetes: Untrained subjects WITH/WITHOUT Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS: Untrained subjects WITH and WITHOUT diabetes used Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood (and study staff tested subject fingerstick blood) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
Period: Overall Study
Arm/Group | Persons With and Without Diabetes
Started | 372
Completed | 372
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The 'Persons With Diabetes' Arm (329) is a subset of the 'Persons With and Without Diabetes' Arm (372).
Groups:
- Persons With and Without Diabetes: Untrained subjects WITH/WITHOUT Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS: Untrained subjects WITH (329) and WITHOUT (43) diabetes used Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood (and study staff tested subject fingerstick blood) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 372
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47
  Not Hispanic or Latino | 320
  Unknown or Not Reported | 5
Race (NIH/OMB) [Number; unit: responses] — Subjects provided more than one choice for Race, therefore the apparent frequency total for Race was different from number of subjects.
  responses
    American Indian or Alaska Native | 7
    Asian | 23
    Native Hawaiian or Other Pacific Islander | 4
    Black or African American | 32
    White | 305
    More than one race | 6
    Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 372

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Untrained subjects WITH diabetes (329) self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 324 (329-5) Blood glucose results were analyzed. One (1) subject had no hematocrit result, required per protocol. For one subject time between subject meter test and collection of subject reference sample exceeded time allowed in protocol. Three subjects did not obtain meter BG result after three attempts.
Measure: Number; unit: Blood glucose results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained subjects WITH Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH (329) Diabetes Use Karajishi Contour BGMS: Untrained subjects WITH diabetes used the Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 324
Blood glucose results within 15mg/dL/15% | 317

2. Secondary Outcome: Number of Venous Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Study staff tested venous blood of subjects WITH diabetes (329) using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results were compared with subject venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer venous plasma BG results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI venous plasma) and +/-15% (>=100 mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 318 (329-11) Blood glucose results were analyzed. Eleven (11) subjects had unsuccessful venipuncture attempts, so no venous results were obtained for them.
Measure: Number; unit: Blood glucose results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained subjects WITH Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH Diabetes Use Karajishi Contour BGMS: Study staff tested subject venous blood from subjects WITH Diabetes (329) and BG results were compared to reference method results obtained from subject venous plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 318
Blood glucose results within 15mg/dL/15% | 318

3. Secondary Outcome: Number of Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method When Obtained and Tested by Study Staff
Description: Study staff obtained and tested subject (329 WITH diabetes) fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 326 (329-3) Blood glucose results were analyzed. One (1) subject had no hematocrit result, required per protocol. One subject had no BG result obtained by study staff. One subject's staff-obtained BG result was not evaluable due to protocol deviation.
Measure: Number; unit: Blood glucose results within 15mg/dL/15%
Groups:
- Persons With Diabetes: Untrained subjects WITH Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH Diabetes Use Karajishi Contour BGMS: Study staff tested subject fingerstick blood (329 WITH Diabetes) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 326
Blood glucose results within 15mg/dL/15% | 325

4. Secondary Outcome: Number of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements
Description: Staff obtained responses from persons WITH diabetes (329) using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' or 'Agree' or 'Neutral' or 'Disagree' or 'Strongly Disagree.'
Time Frame: 1 hour
Measure: Number; unit: number who strongly agree,agree,neutral
Groups:
- Persons With Diabetes: Untrained subjects WITH Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH Diabetes Use Karajishi Contour BGMS: Untrained subjects WITH diabetes (329) used the Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood (and study staff tested subject fingerstick blood) using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
Arm/Group | Persons With Diabetes
Number analyzed (Participants) | 329
number who strongly agree,agree,neutral
  I find it easy to do a blood test with this meter | 326
  The meter display is easy to see and read. | 329
  It was easy to understand my test results. | 329
  I like the overall meter design. | 326
  I find the meter easy to use. | 328
  Instructions (User Guide) were easy to understand. | 326
  Instructions clearly explain how to run a test. | 327
  Instructions clearly explain meter error messages. | 329

5. Secondary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH diabetes (329) and WITHOUT diabetes (43) self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/-15% of the laboratory method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: 365 (372-7) Blood glucose results were analyzed. One (1) subject had no hematocrit result, required per protocol. For one subject time between subject meter test and collection of subject reference sample exceeded time allowed in protocol. Five subjects did not obtain meter BG result after three attempts.
Measure: Number; unit: Blood glucose results within +/- 15%
Groups:
- Persons With and Without Diabetes: Untrained subjects WITH/WITHOUT Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS: Untrained subjects WITH and WITHOUT diabetes used Karajishi Contour BGMS (Blood Glucose Monitoring System). Subjects tested capillary fingerstick blood using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 365
Blood glucose results within +/- 15% | 353

6. Secondary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 20% of Laboratory Glucose Method Across the Tested Glucose Range
Description: Untrained subjects WITH diabetes (329) and WITHOUT diabetes (43) self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/-20% of the laboratory method across the entire tested YSI glucose range.
Time Frame: 1 hour
Population: as for outcome 5
Measure: Number; unit: Blood glucose results within +/- 20%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 365
Blood glucose results within +/- 20% | 359

7. Secondary Outcome: Number of Subject Fingerstick Blood Glucose (BG) Results Within +/- 15% of Laboratory Glucose Method When Obtained and Tested by Study Staff
Description: Study staff obtained and tested subject (WITH and WITHOUT diabetes) fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results were used to calculate the number of BGMS results within +/-15% across the tested YSI glucose range.
Time Frame: 1 hour
Population: 369 (372-3) Blood glucose results were analyzed. One (1) subject had no hematocrit result, required per protocol. For one subject staff test was not performed and for one subject staff test was not evaluable due to protocol deviation.
Measure: Number; unit: Blood glucose results within +/- 20%
Groups:
- Persons With and Without Diabetes: Untrained subjects WITH/WITHOUT Diabetes use Karajishi Contour BGMS (Blood Glucose Monitoring System).
  Subjects WITH/WITHOUT Diabetes Use Karajishi Contour BGMS: Study staff tested subject fingerstick blood using the Karajishi Contour BGMS. All BG results were compared to reference method results obtained with subject capillary plasma.
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 369
Blood glucose results within +/- 20% | 365

8. Secondary Outcome: Number of Subject Fingerstick Blood Glucose (BG) Results Within +/- 20% of Laboratory Glucose Method When Obtained and Tested by Study Staff
Description: Study staff obtained and tested subject (WITH and WITHOUT diabetes) fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results were used to calculate the number of BGMS results within +/-20% across the tested YSI glucose range.
Time Frame: 1 hour
Population: as for outcome 7
Measure: Number; unit: Blood glucose results within +/- 20%
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 369
Blood glucose results within +/- 20% | 367

9. Secondary Outcome: Number of Subject Responses That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements
Description: Staff obtained responses from subjects WITH and WITHOUT diabetes using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' or 'Agree' or 'Neutral' or 'Disagree' or 'Strongly Disagree.'
Time Frame: 1 hour
Measure: Number; unit: Number who strongly agree,agree,neutral
Arm/Group | Persons With and Without Diabetes
Number analyzed (Participants) | 372
Number who strongly agree,agree,neutral
  I find it easy to do a blood test with this meter. | 368
  The meter display is easy to see and read. | 371
  It is easy to understand my test results. | 371
  I like the overall meter design. | 368
  I find the meter easy to use. | 369
  The instruction (User Guide) is easy to understand | 368
  Instructions clearly explain how to run a test. | 368
  Instructions clearly explain meter error messages. | 371

ADVERSE EVENTS:
Arm/Group | Persons With and Without Diabetes
Serious Adverse Events (participants affected / at risk) | 0/372
Other Adverse Events (participants affected / at risk) | 16/372
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persons With and Without Diabetes (N=372)
Hypoglycemia (Endocrine disorders) | 15 (15)
Presyncope (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days